Official Title of Study: Alcohol PBS and Thinking about the Past

**NCT Number:** Not Assigned

Unique Protocol ID: IRB20201070D

**Date of Document:** 09/10/2021

### TEXAS A&M UNIVERSITY HUMAN RESEARCH PROTECTION PROGRAM

#### INFORMED CONSENT

# Title of Research Study: Alcohol Protective Behavioral Strategies and Thinking about the Past

Investigator: Dr. Rachel Smallman

## Why am I being asked to take part in this research study?

You were selected as a possible participant in this study because you are currently enrolled in a psychology course at Texas A&M University. This study is about ways we think about past events, protective behavioral strategies, and alcohol consumption among college students. You must be at least 18 years old, able to speak English fluently, and be able to consent to participate in research. You must also have completed the first part of this study.

# Why is this research being done?

The purpose of this study is to observe the interaction between protective behavioral strategies that college students use and alcohol related problems that may occur while drinking.

# How long will the research last?

There are a total of six parts to this study. Each part will take place exactly one week apart. Each study session will be no more than 30 minutes each.

In the follow up parts of the study, you will be asked to fill out various measures online on alcohol use and alcohol consumption. These follow up sessions will take no more than 30 minutes each. Each follow up session will be one week apart from one another over the span of 5 weeks.

In total, the follow up sessions will take part in five 30-minute sessions over the course of five weeks.

Part 1: Baseline (Previously completed)

Part 2: First follow up (One week after baseline)

Part 3: Second follow up (One week after Part 2)

Part 4: Third follow up (One week after Part 3)

Part 5: Fourth follow up (One week after Part 4)

Part 6: Fifth follow up (One week after Part 5)



#### **INFORMED CONSENT SCRIPT**

# What happens if I say "Yes, I want to be in this research"?

If you decide to participate, please do the following: follow the on-screen computer prompts and instructions. You will complete questionnaires that assess demographic characteristics, alcohol use patterns, alcohol related problems, and protective behavioral strategies. You can skip any question you do not wish to answer, or exit the survey at any point.

## What happens if I do not want to be in this research?

Your participation in this study is voluntary. You can decide not to participate in this research and it will not be held against you. You can leave the study at any time.

# Is there any way being in this study could harm me?

There is a legal risk, as some of these questions ask about alcohol consumption. If you wish to take part in the study, we advise you to do so in a private setting where you feel comfortable about answering such questions.

If at any point you would like to speak with someone about any distress or discomfort you have experienced from the study, please feel free to contact the following resources:

Counseling and Psychological Services: caps.tamu.edu (979)845-4427 Helpline (Crisis Hotline *after hours or after 5 p.m.*): caps.tamu.edu (979)845-2700

There is also a risk of discomfort, as some of the questions are about alcohol use and personal questions about alcohol consumption. You can skip any question you do not wish to answer, or exit the survey at any point.

# What happens to the information collected for the research?

Your *TAMU email address* will be stored separately from your survey data, and is only being collected for the purpose of matching participant data across all parts of the study. All identifiable information will be kept on a password protected server housed within the College of Liberal Arts at Texas A&M University and is only accessible by the research team. Compliance offices at Texas A&M may be given access to the study files upon request.

Your information will be kept confidential to the extent allowed by law. The results of the research study may be published but your identity will remain confidential.

#### **INFORMED CONSENT SCRIPT**

#### What else do I need to know?

You will be granted one research credit to your TAMU SONA account at the end of each part of the study, with a possibility of six total credits earned.

#### Who can I talk to?

Please feel free to ask questions regarding this study. You may contact Dr. Rachel Smallman later if you have additional questions or concerns by phone at 845-3983 or by email at rsmallman@tamu.edu.

You may also contact the Human Research Protection Program at Texas A&M University (which is a group of people who review the research to protect your rights) by phone at 1-979-458-4067, toll free at 1-855-795-8636, or by email at <a href="mailto:irb@tamu.edu">irb@tamu.edu</a> for:

- additional help with any questions about the research
- voicing concerns or complaints about the research
- obtaining answers to questions about your rights as a research participant
- concerns in the event the research staff could not be reached
- the desire to talk to someone other than the research staff

If you want a copy of this consent for your records, you can print it from the screen.

- If you wish to participate, please click the "I Agree" button and you will be taken to the survey.
- If you do not wish to participate in this study, please select "I Disagree" or select X in the corner of your browser